CLINICAL TRIAL: NCT04038944
Title: Anticoagulant and Antiarrhythmic Management Based on Continuous Rhythm Monitoring and Cardiac Imaging in Patients at Low Risk for Cardiovascular Events Following Direct Current Cardioversion for New Onset Atrial Fibrillation
Brief Title: Anticoagulant and Antiarrhythmic Management Based on Continuous Rhythm Monitoring
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: St. Francis Hospital, New York (Other)
Responsible Party: Sponsor
Other Study IDs: 18-19
Record Dates: First submitted 2019-07-29; First posted 2019-07-31 (Actual); Last update posted 2019-07-31 (Actual); Status verified 2019-07

CONDITIONS: New Onset Atrial Fibrillation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Subjects with new onset atrial fibrillation: Subjects with new onset atrial fibrillation who may or may not require electrical cardioversion

SUMMARY:
This pilot study aims to assess the feasibility and safety of using an ILR to identify the incidence of recurrent AF after an episode of newly diagnosed AF. The study further aims to assess the risk of AF recurrence in this low risk population based on left atrial and left atrial appendage anatomic and functional indices in addition to the standardized clinical CHA2DS2-Vasc score.

DETAILED DESCRIPTION:
There is a significant incidence of recurrent AF following initial diagnosis of AF.

Inclusion of left atrial (LA) and left atrial appendage (LAA) abnormalities together with risk prediction of CVA using CHA2DS2-Vasc score will identify patients at low or high risk for adverse cardiovascular events in patients with manifest and silent AF.

Patients requiring cardioversion have higher risk of recurrent AF in follow up.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years
2. Newly diagnosed AF
3. Patient or legal guardian is willing and able to provide informed written consent and comply with follow-up visits and testing schedule

Exclusion Criteria:

1. Patient is participating in or plans to participate in any other investigational drug or device clinical trial that has not reached its primary endpoint
2. Patient received an organ transplant, or is on a waiting list.
3. Patient is not able to follow instructions for remote monitoring 4 Prior history of AF

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The trial will include 250 subjects who have been identified with initial diagnosis of AF and for whom a rhythm control strategy has been chosen with the primary endpoint being time to AF recurrence, AF burden, and AF management at 1 and 3 years.
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2019-07-17 (Actual); Primary Completion 2020-07 (Estimated); Study Completion 2023-09 (Estimated)

PRIMARY OUTCOMES:
Time to AF recurrence | 3 years
  Time to AF recurrence based on clinical or ILR monitoring

SECONDARY OUTCOMES:
All cause death | 30 days; 6 months; 1 year; 2 years; 3 years
  Composite endpoint of all-cause death
AF related re hospitalizations | 3 years
  any hospitalization related to AFib
Occurrence of CVA | 3 years
  Stroke mRs>1 or TIA
Major and minor bleeding | 3 years
  events of major and minor bleeding

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Levine, MD, Principal Investigator — Saint Francis Hospital
Locations (2):
- United States (2):
  - St Francis Hospital, Roslyn, New York
  - St. Francis Hospital, Roslyn, New York

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bai Y, Wang YL, Shantsila A, Lip GYH. The Global Burden of Atrial Fibrillation and Stroke: A Systematic Review of the Clinical Epidemiology of Atrial Fibrillation in Asia. Chest. 2017 Oct;152(4):810-820. doi: 10.1016/j.chest.2017.03.048. Epub 2017 Apr 17. PMID 28427968
- [Background] Staerk L, Sherer JA, Ko D, Benjamin EJ, Helm RH. Atrial Fibrillation: Epidemiology, Pathophysiology, and Clinical Outcomes. Circ Res. 2017 Apr 28;120(9):1501-1517. doi: 10.1161/CIRCRESAHA.117.309732. PMID 28450367
- [Background] Wolf PA, Abbott RD, Kannel WB. Atrial fibrillation as an independent risk factor for stroke: the Framingham Study. Stroke. 1991 Aug;22(8):983-8. doi: 10.1161/01.str.22.8.983. PMID 1866765
- [Background] Hijazi Z, Lindback J, Alexander JH, Hanna M, Held C, Hylek EM, Lopes RD, Oldgren J, Siegbahn A, Stewart RA, White HD, Granger CB, Wallentin L; ARISTOTLE and STABILITY Investigators. The ABC (age, biomarkers, clinical history) stroke risk score: a biomarker-based risk score for predicting stroke in atrial fibrillation. Eur Heart J. 2016 May 21;37(20):1582-90. doi: 10.1093/eurheartj/ehw054. Epub 2016 Feb 25. PMID 26920728
- [Background] Hijazi Z, Oldgren J, Lindback J, Alexander JH, Connolly SJ, Eikelboom JW, Ezekowitz MD, Held C, Hylek EM, Lopes RD, Yusuf S, Granger CB, Siegbahn A, Wallentin L; ARISTOTLE and RE-LY Investigators. A biomarker-based risk score to predict death in patients with atrial fibrillation: the ABC (age, biomarkers, clinical history) death risk score. Eur Heart J. 2018 Feb 7;39(6):477-485. doi: 10.1093/eurheartj/ehx584. PMID 29069359
- [Background] Calenda BW, Fuster V, Halperin JL, Granger CB. Stroke risk assessment in atrial fibrillation: risk factors and markers of atrial myopathy. Nat Rev Cardiol. 2016 Sep;13(9):549-59. doi: 10.1038/nrcardio.2016.106. Epub 2016 Jul 7. PMID 27383079
- [Background] Goldberger JJ, Arora R, Green D, Greenland P, Lee DC, Lloyd-Jones DM, Markl M, Ng J, Shah SJ. Evaluating the Atrial Myopathy Underlying Atrial Fibrillation: Identifying the Arrhythmogenic and Thrombogenic Substrate. Circulation. 2015 Jul 28;132(4):278-91. doi: 10.1161/CIRCULATIONAHA.115.016795. PMID 26216085
- [Background] Andersson T, Magnuson A, Bryngelsson IL, Frobert O, Henriksson KM, Edvardsson N, Poci D. All-cause mortality in 272,186 patients hospitalized with incident atrial fibrillation 1995-2008: a Swedish nationwide long-term case-control study. Eur Heart J. 2013 Apr;34(14):1061-7. doi: 10.1093/eurheartj/ehs469. Epub 2013 Jan 14. PMID 23321349
- [Background] Hart RG, Pearce LA, Aguilar MI. Meta-analysis: antithrombotic therapy to prevent stroke in patients who have nonvalvular atrial fibrillation. Ann Intern Med. 2007 Jun 19;146(12):857-67. doi: 10.7326/0003-4819-146-12-200706190-00007. PMID 17577005
- [Background] Go AS, Hylek EM, Phillips KA, Chang Y, Henault LE, Selby JV, Singer DE. Prevalence of diagnosed atrial fibrillation in adults: national implications for rhythm management and stroke prevention: the AnTicoagulation and Risk Factors in Atrial Fibrillation (ATRIA) Study. JAMA. 2001 May 9;285(18):2370-5. doi: 10.1001/jama.285.18.2370. PMID 11343485
- [Background] European Heart Rhythm Association; European Association for Cardio-Thoracic Surgery; Camm AJ, Kirchhof P, Lip GY, Schotten U, Savelieva I, Ernst S, Van Gelder IC, Al-Attar N, Hindricks G, Prendergast B, Heidbuchel H, Alfieri O, Angelini A, Atar D, Colonna P, De Caterina R, De Sutter J, Goette A, Gorenek B, Heldal M, Hohloser SH, Kolh P, Le Heuzey JY, Ponikowski P, Rutten FH. Guidelines for the management of atrial fibrillation: the Task Force for the Management of Atrial Fibrillation of the European Society of Cardiology (ESC). Eur Heart J. 2010 Oct;31(19):2369-429. doi: 10.1093/eurheartj/ehq278. Epub 2010 Aug 29. No abstract available. PMID 20802247
- [Background] Gage BF, Waterman AD, Shannon W, Boechler M, Rich MW, Radford MJ. Validation of clinical classification schemes for predicting stroke: results from the National Registry of Atrial Fibrillation. JAMA. 2001 Jun 13;285(22):2864-70. doi: 10.1001/jama.285.22.2864. PMID 11401607
- [Background] Hijazi Z, Lindahl B, Oldgren J, Andersson U, Lindback J, Granger CB, Alexander JH, Gersh BJ, Hanna M, Harjola VP, Hylek EM, Lopes RD, Siegbahn A, Wallentin L. Repeated Measurements of Cardiac Biomarkers in Atrial Fibrillation and Validation of the ABC Stroke Score Over Time. J Am Heart Assoc. 2017 Jun 23;6(6):e004851. doi: 10.1161/JAHA.116.004851. PMID 28645934